CLINICAL TRIAL: NCT05361824
Title: Ketorolac Verses Paracetamol as an Adjunct to Nalbuphine in Post Operative Pain Management in Elective Cardiac Surgery
Brief Title: Ketorolac-an Option for Post Operative Pain Management After Elective Cardiac Surgery.
Acronym: KOPAC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Cardiovascular Diseases, Pakistan (Other)
Responsible Party: Principal Investigator, Dr Maaida Muzaffar, Registrar Anesthesia, National Institute of Cardiovascular Diseases, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ERC-83/2020
Record Dates: First submitted 2022-04-30; First posted 2022-05-05 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Coronary Artery Disease; Post Operative Pain; Analgesia; Coronary Artery Bypass Grafting Surgery
MeSH Terms: conditions — Coronary Artery Disease; Pain, Postoperative; Agnosia | interventions — Ketorolac; Ketorolac Tromethamine; Acetaminophen; Valsartan

STUDY DESIGN:
Intervention Model Description: Computer generated, randomized selection of patients with 50% probability of assignment into either group Treatment group : Ketorolac group Control Group: Paracetamol
Who Masked: Participant
Masking Description: 100ml infusion bottles identical in every aspect, except a unique label on them which was only known to investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ketorolac (Experimental): Ketorolac 30mg 8 hourly for 48 hours post-operatively
  Interventions: Drug: Ketorolac Injection
- Paracetamol (Active Comparator): Paracetamol 1gm 6 hourly for 48 hours post-operatively
  Interventions: Drug: Paracetamol

INTERVENTIONS:
Drug: Ketorolac Injection — dosage form: intravenous dosage: 30mg frequency: 8 hours apart (TDS) duration: for 48 hours post operatively
  Other Names: Toradol
  Arms: Ketorolac
Drug: Paracetamol — dosage form: intravenous dosage: 1gm frequency: 6 hours apart (QID) duration: for 48 hours post operatively
  Other Names: Bofalgan; Provas
  Arms: Paracetamol

SUMMARY:
OBJECTIVE: The purpose of this study was to compare the efficacy of Ketorolac versus Paracetamol as an adjunct to Nalbuphine in the management of post-operative pain following elective cardiac surgery.

STUDY DESIGN: Randomized (single-blind) control trial.

SAMPLING TECHNIQUE: Computer generated, randomized selection of patients with 50% probability of assignment into either group.

PLACE AND STUDY DURATION: (single center) SICU at the National Institute of Cardiovascular Diseases Hospital, Karachi over a period of six months, from January 1, 2021 up to June 30, 2021.

METHODS: Sixty patients (30 in each group) were randomly assigned to receive either Paracetamol (control) or Ketorolac (treatment), along with the usual Nalbuphine infusion, over the first 48 hours postoperatively. The control group received injection Paracetamol 1gm six hourly, whereas treatment group received injection Ketorolac 30mg eight hourly.

PRIMARY OUTCOME: The VAS (pain score) was evaluated at 6, 12, 18 and 24 hours post-extubation and a score of 4 or less was taken as a cut-off for adequate pain control.

SECONDARY OUTCOMES: The time taken to extubation postoperatively. The total dose of Nalbuphine administered to each patient and total chest tube drainage recorded over 48 hours postoperatively.

DETAILED DESCRIPTION:
DATA COLLECTION: Computer randomization was done for the numbers 1 to 60, having 50% probability of being in either of two groups: Ketorolac (treatment) or Paracetamol (control).

After randomizing each number into either group, which ever patient (consenting and meeting the inclusion criteria) came, was allotted these numbers consecutively, as they presented for elective cardiac surgery. Thus randomly allocating the presenting patients into either Ketorolac/treatment (30 patients) and Paracetamol/control (30 patients).

Each patient was explained about the VAS pain rating score twice; first at preoperative interview and second time after they recovered their alert state in the SICU post operatively( at time of extubation).

The patients were taught to finger-point their intensity of pain on a line between two endpoints: marked 0 to 10. Mark at '0' meant no pain at all and '10' worst pain ever felt. The number that the patient pointed to, defined the patient's pain. For the purposes of this study "adequate pain relief" was defined as achieving a pain score of four or less, this designation was also included on the VAS scale and explained to the patients so that they may indicate numbers higher than four if they felt any pain.

Standard anaesthesia was given in the operative room, total analgesia given intra-operatively was 0.4 mg/kg Nalbuphine (not exceeding 30mg).

After completion of the surgery all patients were shifted to SICU. Initially both groups received a bolus dose of 10mg Nalbuphine and then an infusion of Nalbuphine was started at 2.5mg/hr as maintenance, up to 24 hours post-operatively. In addition, (according to randomization) the patients in treatment group received Ketorolac 30mg 8 hourly for 48 hours post-operatively and the patients control group received Paracetamol 1gm 6 hourly for 48 hours post-operatively.

Postoperative analgesia assessment using VAS was performed at 6 hours, 12 hours, 18 hours and 24 hours postextubation.

Time taken to extubation, total dose of Nalbuphine administered to each patient and total chest tube drainage were also recorded over 24 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 18 years and above of age.
* Undergoing elective cardiac surgery.
* American Society of Anesthesiology (ASA) Physical Class 3 or 4.

Exclusion Criteria:

* • Patients pre-planned for delayed extubation (due to moderate to severe pulmonary artery hypertension, poor right ventricular function, rhythm disturbances or unstable vitals)

  * Low cardiac output (cardiac index < 2.0 l/min/m2, using transesophageal echocardiography, intraoperatively) after weaning off cardiopulmonary bypass or paitients already having pre-op ejection fraction < 30%.
  * Patients not comfortably ventilated or oxygenated, requiring high doses of sedation and neuromuscular blockage.
  * Sensitivity or allergy to nonsteroidal anti-inflammatory drugs.
  * History of peptic ulcer or gastrointestinal bleeding.
  * Serum creatinine = 2.0 mg/dl or increase in serum creatinine of = 0.5 mg/dl or 25% within the preceding 10 days.
  * Hepatic dysfunction.
  * Bleeding disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-06 (Actual)

PRIMARY OUTCOMES:
Reduction in pain severity | 6 hours apart for total 24 hours(6 hours, 12 hours , 18 hours and 24 hours) post extubation.
  Post operative analgesic assessment using Visual Analogue Scale VAS: a 10 cm long line between the two endpoints (0 to 10). 0: no pain at all 10: worst pain ever felt The mark that the patient pointed to, defined the patient's pain. For the purposes of this study "adequate pain relief" was defined as achieving a pain score of four or less, this designation was also included on the VAS scale and explained to the patients so that they may indicate numbers higher than four if they felt any pain.

SECONDARY OUTCOMES:
Reduction in Opioid usage (if any) | Within 48 hours postoperatively
  Reduction in Nalbuphine administration as an opioid analgesic
Time to Extubation in hours | Within 24 hours postoperatively
  Time taken from patient's entry into the surgical ICU after elective cardiac surgery, till the time Endotracheal tube was removed.
Total amount of blood (in milliliters) collected, in the under-water sealed drain bottles, via chest drainage tubes | Within 48 hours postoperatively
  The total amount (in milliliters) of blood collected via chest drains into the under-water sealed drain bottles

CONTACTS AND LOCATIONS:
Overall Officials: Dr Maaida Muzaffar, FCPS, Principal Investigator — National Institute of Cardiovascular Diseases, Pakistan
Locations (1):
- National Institute of Cardiovascular Diseases, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
Only patient's unique hospital ID will be provided if required